CLINICAL TRIAL: NCT02628392
Title: A Phase 2, Randomized, Double-blind, Dose Finding Study of DS-8500a in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: A Phase 2 Study of DS-8500a in Japanese Subjects With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS8500-A-J203
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2017-01

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Adult; Developmental Phase II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — firuglipel; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- DS-8500a 25 mg QD (Experimental): DS-8500a 25 mg tablet once daily (QD), orally, for up to 12 weeks, and matching sitagliptin placebo capsule
  Interventions: Drug: DS-8500a; Drug: placebo
- DS-8500a 50 mg QD (Experimental): DS-8500a 50 mg QD tablet, orally, once daily for up to 12 weeks, and matching sitagliptin placebo capsule
  Interventions: Drug: DS-8500a; Drug: placebo
- DS-8500a 75 mg QD (Experimental): DS-8500a 75 mg QD tablet, orally, once daily for up to 12 weeks, and matching sitagliptin placebo capsule
  Interventions: Drug: DS-8500a; Drug: placebo
- placebo (Placebo Comparator): placebo tablet and placebo capsule, orally, once daily for up to 12 weeks to match DS-8500a and sitagliptin, respectively.
  Interventions: Drug: placebo
- Sitagliptin (Active Comparator): capsule, orally, once daily for up to 12 weeks and matching DS-8500 placebo tablet
  Interventions: Drug: Sitagliptin; Drug: placebo

INTERVENTIONS:
Drug: DS-8500a — DS-8500a tablets 25mg, 50mg, 75mg
  Arms: DS-8500a 25 mg QD; DS-8500a 50 mg QD; DS-8500a 75 mg QD
Drug: Sitagliptin — capsules
  Other Names: Januvia
  Arms: Sitagliptin
Drug: placebo — matching DS-8500a tablets and sitagliptin capsules

SUMMARY:
The objectives of the study is to evaluate the efficacy, safety, and dose of DS-8500a compared with placebo in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The objectives of the study is to evaluate the efficacy, safety, and dose of DS-8500a compared with placebo in patients with type 2 diabetes mellitus after a 12-week oral administration of DS-8500a at 25, 50, or 75 mg in a double-blind, parallel-group comparison study. In addition, the clinical positioning of DS-8500a relative to an existing drug will be investigated using sitagliptin as a comparator.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 20 years at the time of informed consent
* Japanese patients with type 2 diabetes
* Patients who have HbA1c ≥ 7.0% and < 10.0%

Exclusion Criteria:

* Patients with type 1 diabetes mellitus or with a history of diabetic coma, precoma, or ketoacidosis
* Patients receiving or requiring treatment with insulin
* Patients with a body mass index (BMI) of < 18.5 kg/m2 or ≥ 35.0 kg/m2
* Patients with clinically evident renal impairment (estimated glomerular filtration rate [eGFR] of < 45 mL/min per 1.73 m2) or clinically significant renal disease
* Patients with fasting plasma glucose ≥ 240 mg/dL

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
change in HbA1c | baseline (Day -1) to Week 12
  HbA1c = glycated hemoglobin

SECONDARY OUTCOMES:
change in HbA1c | baseline (Day -1) to Week 4
change in HbA1c | baseline (Day -1) to Week 8
proportion of subjects with HbA1c <7.0 | baseline (Day -1) to Week 12
  proportion of subjects who achieve HbA1c <7.0
change in plasma glucose | baseline (Day -1) to Week 4
change in plasma glucose | baseline (Day -1) to Week 12
change in AUC derived from plasma glucose | baseline (Day -1) to Week 4
  change in pharmacodynamics profile consists of Area Under Curve (AUC), Concentration maximum (Cmax), Time of maximum concentration (Tmax)
change in AUC derived from plasma glucose | baseline (Day -1) to Week 12
  pharmacodynamics profile consists of AUC, Cmax, Tmax
change in serum insulin | baseline (Day -1) to Week 4
change in AUC 0-3h serum insulin | baseline (Day -1) to Week 4
change in serum insulin | baseline (Day -1) to Week 12
change in AUC 0-3h serum insulin | baseline (Day -1) to Week 12
change in proinsulin | baseline (Day -1) to Week 4
change in AUC 0-3h proinsulin | baseline (Day -1) to Week 4
change in proinsulin | baseline (Day -1) to Week 12
change in AUC 0-3h proinsulin | baseline (Day -1) to Week 12
change in C-peptide | baseline (Day -1) to Week 4
change in AUC 0-3h C-peptide | baseline (Day -1) to Week 4
change in C-peptide | baseline (Day -1) to Week 12
change in AUC 0-3h C-peptide | baseline (Day -1) to Week 12
change in PYY | baseline (Day -1) to Week 4
  PYY = peptide YY
change in AUC 0-3h PYY | baseline (Day -1) to Week 4
change in PYY | baseline (Day -1) to Week 12
change in AUC 0-3h PYY | baseline (Day -1) to Week 12
change in total GLP-1 | baseline (Day -1) to Week 4
  GLP-1 = Glucagon-Like Peptide-1
change in total AUC 0-3h GLP-1 | baseline (Day -1) to Week 4
change in total GLP-1 | baseline (Day -1) to Week 12
change in AUC 0-3h total GLP-1 | baseline (Day -1) to Week 12
change in active GLP-1 | baseline (Day -1) to Week 4
change in AUC 0-3h active GLP-1 | baseline (Day -1) to Week 4
change in active GLP-1 | baseline (Day -1) to Week 12
change in AUC 0-3h active GLP-1 | baseline (Day -1) to Week 12
change in total GIP | baseline (Day -1) to Week 4
  GIP = Gastric Inhibitory Polypeptide
change in AUC 0-3h total GIP | baseline (Day -1) to Week 4
change in total GIP | baseline (Day -1) to Week 12
change in AUC 0-3h total GIP | baseline (Day -1) to Week 12
change in glucagon | baseline (Day -1) to Week 4
change in AUC 0-3h glucagon | baseline (Day -1) to Week 4
change in glucagon | baseline (Day -1) to Week 12
change in AUC 0-3h glucagon | baseline (Day -1) to Week 12
change in 1,5 AG | baseline (Day -1) to Week 4
  1,5 AG = 1,5 anhydrogucitol
change in AUC 0-3h 1,5 AG | baseline (Day -1) to Week 4
change in 1,5 AG | baseline (Day -1) to Week 12
change in AUC 0-3h 1,5 AG | baseline (Day -1) to Week 12
change in total cholesterol | baseline (Day -1) to Week 2
change in total cholesterol | baseline (Day -1) to Week 4
change in total cholesterol | baseline (Day -1) to Week 8
change in total cholesterol | baseline (Day -1) to Week 12
change in HDL cholesterol | baseline (Day -1) to Week 2
  HDL = high density lipoprotein
change in HDL cholesterol | baseline (Day -1) to Week 4
change in HDL cholesterol | baseline (Day -1) to Week 8
change in HDL cholesterol | baseline (Day -1) to Week 12
change in LDL cholesterol | baseline (Day -1) to Week 2
  LDL = low density lipoprotein
change in LDL cholesterol | baseline (Day -1) to Week 4
change in LDL cholesterol | baseline (Day -1) to Week 8
change in LDL cholesterol | baseline (Day -1) to Week 12
change in triglyceride | baseline (Day -1) to Week 2
change in triglyceride | baseline (Day -1) to Week 4
change in triglyceride | baseline (Day -1) to Week 8
change in triglyceride | baseline (Day -1) to Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Heishinkai Medical Group Incorporated OCROM Clinic, Suita-shi, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/